CLINICAL TRIAL: NCT06186726
Title: Prospective Phase II Clinical Study of Carbon Ion Radiotherapy Combined With Chemotherapy for Thymic Epithelial Tumors
Brief Title: Clinical Study of Carbon Ion Radiotherapy Combined With Chemotherapy for Thymic Epithelial Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jian Chen (Other)
Responsible Party: Sponsor-Investigator, Jian Chen, Clinical Professor, Shanghai Proton and Heavy Ion Center
Organization: Shanghai Proton and Heavy Ion Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-THLC2023-04
Record Dates: First submitted 2023-12-17; First posted 2024-01-02 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Carbon Ion Radiotherapy, Thymoma, Thymic Carcinoma, Radiotherapy, Chemotherapy
MeSH Terms: conditions — Thymoma | interventions — Heavy Ion Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study arm (Experimental): The patients received 72GyE/18 fractions of carbon ion radiotherapy. Combined with platinum-containing schemes (including etoposide combined with cisplatin or carboplatin or loplatin or nedaplatin, paclitaxel combined with cisplatin or carboplatin or loplatin or nedaplatin, etc.); Docetaxel combined with cisplatin or carboplatin or loplatin or nedaplatin) for at least 4 cycles
  Interventions: Radiation: carbon ion radiotherapy

INTERVENTIONS:
Radiation: carbon ion radiotherapy — The patients received 72GyE/18 doses of carbon ion radiotherapy.

SUMMARY:
To observe the efficacy of carbon ion radiotherapy combined with chemotherapy in the treatment of inoperable locally advanced or advanced (all visible lesions can be included in the radiation target area in this treatment) primary thymic epithelial tumor who have no thorax radiotherapy histroy. The patients will receive 72GyE/18fractions of carbon ion radiotherapy. Combined with platinum-containing schemes (including etoposide combined with cisplatin or carboplatin or loplatin or nedaplatin, paclitaxel combined with cisplatin or carboplatin or loplatin or nedaplatin, etc.); Docetaxel combined with cisplatin or carboplatin or loplatin or nedaplatin) for at least 4 cycles. Progression-free survival, local control rate, overall survival and toxicity were calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inoperable locally advanced or advanced thymic epithelial tumor who have been confirmed pathologically, and have not received thoracic radiation therapy before coming to our hospital, and have radiologically evaluable lesions, and all visible lesions can be included in the radiation target area during this treatment.
* Between the ages of 18 and 70.
* Sign the informed consent.
* ECOG general status score of 0-2 .
* The expected survival is greater than or equal to 6 months.
* Adequate organ function: 1). Blood function: absolute neutrophil count (ANC) ≥1.5 x 109/L, platelet count ≥80 x 109/L, hemoglobin ≥9 g/dL 2). Lung function: FEV1>25%, DLCO>25% 3). Cardiac function: no serious pulmonary hypertension, cardiovascular and cerebrovascular diseases, peripheral vascular diseases, serious chronic heart disease and other complications that may affect radiotherapy.4). Adequate liver function: total bilirubin <1.5 times the upper limit of normal value, and AST, ALT<2 times the upper limit of normal value. 5). Adequate renal function: serum creatinine ≤1.5 times the upper limit of normal or calculated creatinine clearance ≥50 ml /min, and urinary protein <2+. Patients with a baseline urinary protein level of 2+ or more should have a 24-hour urine collection and evidence of a 24-hour urinary protein level of 1g or less.

Exclusion Criteria:

* Complicated with other malignant tumors that have not been controlled.
* With large quantity of pleural effusion or pericardial effusion.
* Patient whose particle radiotherapy plan cannot meet the minimum target dose coverage and dose volume limitation requirements, or cannot meet the dose constrains of normal tissue or organs.
* Chest radiation therapy or radioactive particle implantation history.
* Cardiac pacemakers or other internal metal prosthesis implants that may be affected by high-energy radiation or may affect the dose distribution to the radiation target area.
* Pregnancy (confirmed by serum or urine β-HCG test) or lactation period.
* HIV positive. Hepatitis virus replication phase, need to receive antiviral therapy, but because of concomitant disease cannot receive antiviral therapy. Active stage of syphilis.
* A history of mental illness may hinder the completion of treatment.
* With serious comorbidity that may interfere with radiotherapy, including: (a) Acute infectious diseases or acute active phase of chronic infection. b) Unstable angina pectoris, congestive heart failure, myocardial infarction that has been hospitalized in the past 6 months. c) Exacerbations of chronic obstructive pulmonary disease or other respiratory conditions requiring hospitalization. d) Severely impaired immune function. e) Diseases with excessive sensitivity to radiation such as ataxia telangiectasia. f) Other diseases that may affect particle radiotherapy.
* Other circumstances that the physician considers inappropriate to participate in clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease progression-free survival rate | From date of radiotherapy started until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Disease progression-free survival rate was defined from the start of carbon ion radiotherapy till the date of disease progression at any site or death, or the last follow up

SECONDARY OUTCOMES:
Local control rate | From date of radiotherapy started until the date of first documented local disease progression, assessed up to 100 months
  Local control rate was defined from the start of carbon ion radiotherapy till the date of local failure or the last follow-up.
Overall survival rate | From date of radiotherapy started until the date of death from any cause, assessed up to 100 months.
  Overall survival rate was defined from the start of carbon ion radiotherapy till the date of death or the last follow-up.
Incidence of Treatment-induced Adverse Events | From date of radiotherapy started, every 3-4 months within the first 2 years, every 6 months between years 3 and 5, and annually thereafter, assessed up to 100 months.
  Treatment-induced toxicities were scored using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, for events observed after the first dose of irradiation. Toxicities occurred 90 or more days after the completion of CIRT were defined as late toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Chen, M.D., Principal Investigator — Shanghai Proton and Heavy Ion Center
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided